CLINICAL TRIAL: NCT03026439
Title: The Boundaries of Mild Chronic Obstructive Pulmonary Disease: Searching Clinical COPD Onset
Brief Title: Searching Clinical Chronic Obstructive Pulmonary Disease Onset
Acronym: SOON
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 13-125b; 1141108 (Other Grant/Funding Number: FONDECYT)
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Copd
Keywords: mild COPD; early COPD; six-min walk test; computed tomography; emphysema; airway disease; peripheral muscle mass; Saint George's Respiratory Questionnaire
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Non-dyspneic smokers/ normal spirometry: Male or female current or former smokers. Forced expiratory volume in 1 s (FEV1)/forced vital capacity (FVC) >0.7. FVC >lower limit of normal (LLN). Modified Medical Research Council (mMRC) dyspnea score = 0.
- Dyspneic smokers/ normal spirometry: Male or female current or former smokers. FEV1/FVC >0.7. FVC >LLN. mMRC dyspnea score ≥1.
- Non-dyspneic mild COPD patients: Male or female current or former smokers. FEV1/FVC ≤0.7. FEV1 >80% of predicted value. mMRC dyspnea score =0.
- Dyspneic mild COPD patients: Male or female current or former smokers. FEV1/FVC ≤0.7. FEV1 >80% of predicted value. mMRC dyspnea score ≥1.

SUMMARY:
The aim of this study is to determine if presence of dyspnea identifies differences in the 6-min walk test performance among smokers with normal or mild spirometric obstruction, accounting for the confounding effect of heart failure on dyspnea with stress echocardiography.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) has a prolonged course before onset, following classical epidemiological principles of chronic disease and genetic predisposition. "Disease onset" may be defined as a physiologic impairment expressed by an abnormal spirometric index, but "early disease" could include clinical manifestations, such as cough, phlegm, dyspnea or exercise limitation, but normal spirometry. For the present proposal, we will use dyspnea to define a symptomatic subject, since dyspnea is the most relevant symptom all over the range of the disease. Besides, we have defined "early disease" when current or ex-smoker-adults: a) complain of dyspnea but have normal spirometry; b) complain of dyspnea and have mild bronchial obstruction; and, c) have mild bronchial obstruction without dyspnea. These subtypes are roughly similar to Global initiative for Chronic Obstructive Lung Disease (GOLD) stages 0 and 1 [1], although further characterized by the presence or absence of dyspnea. The dyspnea cut off value we have chosen to separate symptomatic from asymptomatic subjects is a modified Medical Research Council (mMRC) score ≥1, which is in line with several recent communications [2-4], but differs from the cut off recommended by GOLD (score ≥2) [5]. In addition, GOLD 0 stage [1], included in the GOLD guidelines of 2001 and currently not in use, did not comprise a dyspneic subtype, which is now included in light of new evidence pointing out at their potential relevance [6, 7].

Early disease subtypes

1. Symptomatic current or ex-smokers with normal spirometry have been reported by Woodruff et al [7] on a large sample of individuals who complain of chronic respiratory symptoms, reduced exercise tolerance, and computed tomography (CT) imaging bronchiolitis. These results are in line with previous findings of another large study from Regan et al [8] where more than 50% of symptomatic smokers with normal spirometry have respiratory-related impairment and evidence of emphysema on CT imaging. Woodruff et al [7] used the COPD Assessment Test (CAT) questionnaire to define symptoms [9] and found that cough, phlegm, dyspnea, activity limitation, and energy level were equally distributed among symptomatic smokers regardless of the presence of spirometric COPD. However, although CAT is intended to be specific for COPD [9], most of its domains may reflect concomitant respiratory (asthma and bronchiectasis) and/or nonrespiratory diseases (heart failure, ischemic heart disease, obesity, and depression) [10]. In contrast, Regan et al [8] measured seven "respiratory-related impairments" and found one or more to be present in 54% of patients. Three of these impairments could be considered rather specific of COPD, like CT percentage of emphysema >5% and gas trapping >20%, and St. George's Respiratory Questionnaire (SGRQ) total score >25. However, four impairments (chronic bronchitis, modified Medical Research Council (mMRC) dyspnea score ≥2, exacerbations and 6-min walk distance <350 m) are non-specific as they may be partly or fully explained by comorbidities like gastroesophageal reflux disease, rhinosinusitis, obesity or heart failure, among others. Actually, retrospective data suggest that patients with COPD and comorbid conditions may have greater risk for having symptoms than those without comorbidity [11, 12].
2. Non-dyspneic current or ex-smokers with mild COPD has been also described [13, 14]. It seems that in this group coexist individuals with normal lung function and 6-min walk test performance [14] and subjects with resting lung hyperinflation, reduced diffusion capacity of the lung for carbon monoxide (DLCO) and slightly increased cycle-exercise-induced dyspnoea [13].
3. Dyspneic current or ex-smokers with mild COPD have significant emphysema and airway thickness, lower DLCO, exercise-induced arterial desaturation, and reduced 6-min walking distance [14, 15]. In addition, during incremental cycle-exercise they exhibit increased ventilatory demand, lung hyperinflation and greater exertional dyspnea than smoker controls [16].

Hypothesis

We hypothesize that dyspneic individuals notwithstanding of their spirometry results, should share some clinical, structural and physiologic abnormalities. In particular, we expect that the two dyspneic groups with and without mild COPD exhibit reduced exercise capacity, in addition to worse quality of life; lower physical activity; greater lung hyperinflation; greater emphysema and airway thickness; and reduced peripheral muscle mass, than their asymptomatic counterpart, i.e., non-dyspneic mild COPD and controls.

Study aim

This study intends to identify the three early COPD subtypes already defined using differences in exercise capacity as the primary outcome. As secondary outcomes, we will intend to separate these groups by means of differences in clinical (quality of life, physical activity), physiological (exercise testing) and structural characteristics (emphysema, airway disease, and peripheral muscle mass by CT imaging). Future analyses are planned to evaluate longitudinal deterioration in these clinical, physiological and structural characteristics. Potential influence of obesity and undiagnosed heart failure on dyspnea and thus, on exercise capacity, will be explored within the three subtypes.

Study design

The study has a cross sectional design aimed at obtaining representative samples of adults between 45 and 80 years. Two hundred and forty participants will be enrolled into four strata as already defined, i.e., dyspneic current or ex-smokers with and without mild COPD; and non-dyspneic current or ex-smokers with and without (controls) mild COPD. Study subjects will be recruited from the outpatient clinics and the pulmonary function labs at the Pontifical Catholic University of Chile Health Network by means of physician referral, advertisement in clinical areas, or self-referral at the study center. The Institutional Ethics Committee approved the study protocol and signed informed consent will be obtained from all participants.

Sample size

A sample size of at least 52 subjects per group provide enough power (80%) to detect a significant difference (95% confidence level or alpha 0.05) in the 6-min walk test among symptomatic and asymptomatic participants, based on a conservative relevant difference in walking distance of 50 meters with a common standard deviation of 110 metres. Such difference was found when comparing symptomatic and asymptomatic subjects with normal spirometry [7], but may be an underestimation in patients with mild spirometric COPD [14], where the difference between symptomatic and asymptomatic patients was 100 metres. Forestalling a participant loss rate of 20%, 60 patients will be included in each group.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 to 80 years
* Smoking history >10 pack-year
* Mild COPD subjects: Male or female individuals; post-bronchodilator forced expiratory volume in 1 s (FEV1) ≥80% of predicted normal and post-bronchodilator FEV1/forced vital capacity (FVC) ratio <0.70
* Non-COPD subjects: Male or female individuals; post-bronchodilator FEV1 ≥80% of predicted normal and post-bronchodilator FEV1/FVC ratio ≥0.70

Exclusion Criteria:

* Unable to tolerate study procedures
* Unable to walk or cycle without assistance
* Dementia or cognitive disorder, which would prevent the participant from consenting the study or completing study procedures
* Major depressive disorder
* Locomotor disease that seriously limits exercise tolerance
* Untreated symptomatic peripheral artery disease
* Body Mass Index >40 kg/m2
* Non-COPD significant pulmonary disease such as asthma; interstitial lung disease; sarcoidosis; tuberculosis; cystic fibrosis; diffuse bronchiectasis; and others
* Primary pulmonary hypertension
* Current lung cancer
* Previous lung resection
* Large thoracic metal implants that in opinion of the investigator limit CT scan analyses
* Current use of prednisone >5 mg daily
* Current use of immunosuppressive agent
* Current exposure to chemotherapy or radiation treatments that, in the opinion of the investigator could limit interpretation of pulmonary function, exercise tolerance and CT scan imaging
* Current illicit substance abuse, excluding marijuana
* Known HIV/AIDS infection
* Current extra thoracic cancer, which, in the opinion of their physicians, limits life expectancy to less than 3 years
* Recent myocardial infarction (6 months or less)
* Chronic congestive heart failure

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects will be recruited from the outpatient clinics and the pulmonary function labs at the Pontifical Catholic University of Chile Health Network by means of physician referral, advertisement in clinical areas, or self-referral at the study centre.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Walking distance during the six-minute walking test | Baseline

SECONDARY OUTCOMES:
Health related quality of life | Baseline
  St. George's Respiratory Questionnaire
Computed tomography emphysema | Baseline
  Emphysema will be quantitated using the percentage of low-attenuation units less than -950 Hounsfield units (HU) using open source software (www.Slicer.org).
Computed tomography airway thickness | Baseline
  Single-slice airway measurements will be collected in the apical bronchus of the right upper lobe and the right lower lobe posterior basal bronchus. Measurements will be performed in the 3rd, 4th, and 5th airway generation.
Computed tomography cross-sectional area of the right thigh muscle | Baseline
  The cross-sectional area of the right thigh muscle will be measured at halfway between the pubic symphysis and the inferior condyle of the femur, in the surface area of the tissue with a density of 40 to 100 HU. This range of density corresponds to the density of muscle tissue.
Lung function | Baseline
  Spirometry, single-breath DLCO, and plethysmographic lung volume assessment will be performed
Stress echocardiography | Baseline
  Transthoracic stress echocardiography will be performed with a VIVID-7 echocardiography system and echo cardiac stress table, with electrical adjustable slope for an optimal position of the heart. Function in each segment of the left ventricle (LV) will be graded at rest and with stress as normal or hyperdynamic, hypokinetic, akinetic, dyskinetic, or aneurysmal. In addition to the evaluation of segmental function, the global LV response to stress be assessed. Diastolic function will be analysed at rest, and systolic function at rest and end exercise
Physical activity | Baseline
  A triaxial accelerometer will be used. This accelerometer measures activity counts and vector magnitude, energy expenditure, steps taken, physical activity intensity, subject position, and ambient light levels. We will retrieve, collect and study three physical activity (PA) outcomes: step count (i.e. movement); spent physical activity time per day (i.e., moderate or vigorous), and PA level (i.e., activity related energy expenditure).
Exercise testing | Baseline
  A symptom-limited incremental cycle exercise test will be conducted to measure the maximal workload. A constant work rate cycle endurance test will be performed afterwards.

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Diaz, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Respiratory Department; Hospital Clinico Universidad Catolica, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pauwels RA, Buist AS, Calverley PM, Jenkins CR, Hurd SS; GOLD Scientific Committee. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease. NHLBI/WHO Global Initiative for Chronic Obstructive Lung Disease (GOLD) Workshop summary. Am J Respir Crit Care Med. 2001 Apr;163(5):1256-76. doi: 10.1164/ajrccm.163.5.2101039. No abstract available. PMID 11316667
- [Background] Han MK, Muellerova H, Curran-Everett D, Dransfield MT, Washko GR, Regan EA, Bowler RP, Beaty TH, Hokanson JE, Lynch DA, Jones PW, Anzueto A, Martinez FJ, Crapo JD, Silverman EK, Make BJ. GOLD 2011 disease severity classification in COPDGene: a prospective cohort study. Lancet Respir Med. 2013 Mar;1(1):43-50. doi: 10.1016/S2213-2600(12)70044-9. Epub 2012 Sep 3. PMID 24321803
- [Background] Jones PW, Adamek L, Nadeau G, Banik N. Comparisons of health status scores with MRC grades in COPD: implications for the GOLD 2011 classification. Eur Respir J. 2013 Sep;42(3):647-54. doi: 10.1183/09031936.00125612. Epub 2012 Dec 20. PMID 23258783
- [Background] Kim S, Oh J, Kim YI, Ban HJ, Kwon YS, Oh IJ, Kim KS, Kim YC, Lim SC. Differences in classification of COPD group using COPD assessment test (CAT) or modified Medical Research Council (mMRC) dyspnea scores: a cross-sectional analyses. BMC Pulm Med. 2013 Jun 3;13:35. doi: 10.1186/1471-2466-13-35. PMID 23731868
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Oelsner EC, Hoffman EA, Folsom AR, Carr JJ, Enright PL, Kawut SM, Kronmal R, Lederer D, Lima JA, Lovasi GS, Shea S, Barr RG. Association between emphysema-like lung on cardiac computed tomography and mortality in persons without airflow obstruction: a cohort study. Ann Intern Med. 2014 Dec 16;161(12):863-73. doi: 10.7326/M13-2570. PMID 25506855
- [Background] Woodruff PG, Barr RG, Bleecker E, Christenson SA, Couper D, Curtis JL, Gouskova NA, Hansel NN, Hoffman EA, Kanner RE, Kleerup E, Lazarus SC, Martinez FJ, Paine R 3rd, Rennard S, Tashkin DP, Han MK; SPIROMICS Research Group. Clinical Significance of Symptoms in Smokers with Preserved Pulmonary Function. N Engl J Med. 2016 May 12;374(19):1811-21. doi: 10.1056/NEJMoa1505971. PMID 27168432
- [Background] Regan EA, Lynch DA, Curran-Everett D, Curtis JL, Austin JH, Grenier PA, Kauczor HU, Bailey WC, DeMeo DL, Casaburi RH, Friedman P, Van Beek EJ, Hokanson JE, Bowler RP, Beaty TH, Washko GR, Han MK, Kim V, Kim SS, Yagihashi K, Washington L, McEvoy CE, Tanner C, Mannino DM, Make BJ, Silverman EK, Crapo JD; Genetic Epidemiology of COPD (COPDGene) Investigators. Clinical and Radiologic Disease in Smokers With Normal Spirometry. JAMA Intern Med. 2015 Sep;175(9):1539-49. doi: 10.1001/jamainternmed.2015.2735. PMID 26098755
- [Background] Karloh M, Fleig Mayer A, Maurici R, Pizzichini MMM, Jones PW, Pizzichini E. The COPD Assessment Test: What Do We Know So Far?: A Systematic Review and Meta-Analysis About Clinical Outcomes Prediction and Classification of Patients Into GOLD Stages. Chest. 2016 Feb;149(2):413-425. doi: 10.1378/chest.15-1752. Epub 2016 Jan 12. PMID 26513112
- [Background] Fabbri LM. Smoking, Not COPD, as the Disease. N Engl J Med. 2016 May 12;374(19):1885-6. doi: 10.1056/NEJMe1515508. No abstract available. PMID 27168438
- [Background] Agusti A, Edwards LD, Celli B, Macnee W, Calverley PM, Mullerova H, Lomas DA, Wouters E, Bakke P, Rennard S, Crim C, Miller BE, Coxson HO, Yates JC, Tal-Singer R, Vestbo J; ECLIPSE Investigators. Characteristics, stability and outcomes of the 2011 GOLD COPD groups in the ECLIPSE cohort. Eur Respir J. 2013 Sep;42(3):636-46. doi: 10.1183/09031936.00195212. Epub 2013 Jun 13. PMID 23766334
- [Background] Agusti A, Hurd S, Jones P, Fabbri LM, Martinez F, Vogelmeier C, Vestbo J, Rodriguez-Roisin R. FAQs about the GOLD 2011 assessment proposal of COPD: a comparative analysis of four different cohorts. Eur Respir J. 2013 Nov;42(5):1391-401. doi: 10.1183/09031936.00036513. Epub 2013 May 3. PMID 23645406
- [Background] Soumagne T, Laveneziana P, Veil-Picard M, Guillien A, Claude F, Puyraveau M, Annesi-Maesano I, Roche N, Dalphin JC, Degano B. Asymptomatic subjects with airway obstruction have significant impairment at exercise. Thorax. 2016 Sep;71(9):804-11. doi: 10.1136/thoraxjnl-2015-207953. Epub 2016 May 25. PMID 27226423
- [Background] Diaz AA, Morales A, Diaz JC, Ramos C, Klaassen J, Saldias F, Aravena C, Diaz R, Lisboa C, Washko GR, Diaz O. CT and physiologic determinants of dyspnea and exercise capacity during the six-minute walk test in mild COPD. Respir Med. 2013 Apr;107(4):570-9. doi: 10.1016/j.rmed.2012.12.011. Epub 2013 Jan 9. PMID 23313036
- [Background] Kirby M, Owrangi A, Svenningsen S, Wheatley A, Coxson HO, Paterson NA, McCormack DG, Parraga G. On the role of abnormal DL(CO) in ex-smokers without airflow limitation: symptoms, exercise capacity and hyperpolarised helium-3 MRI. Thorax. 2013 Aug;68(8):752-9. doi: 10.1136/thoraxjnl-2012-203108. Epub 2013 Apr 19. PMID 23604381
- [Background] Ofir D, Laveneziana P, Webb KA, Lam YM, O'Donnell DE. Mechanisms of dyspnea during cycle exercise in symptomatic patients with GOLD stage I chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Mar 15;177(6):622-9. doi: 10.1164/rccm.200707-1064OC. Epub 2007 Nov 15. PMID 18006885
- [Derived] Labarca G, Bustamante A, Valdivia G, Diaz R, Huete A, Mac Nab P, Mendoza L, Leppe J, Lisboa C, Saldias F, Diaz O. The boundaries of mild chronic obstructive pulmonary disease (COPD): design of the searching clinical COPD onset (SOON) study. BMJ Open. 2017 Aug 11;7(8):e015731. doi: 10.1136/bmjopen-2016-015731. PMID 28801407